CLINICAL TRIAL: NCT03185572
Title: The Prevalence, Disease Course, Prognosis and Interaction of Chronic Obstructive Pulmonary Disease With Pulmonary Hypertension
Brief Title: Registry for Chronic Obstructive Pulmonary Disease With Pulmonary Hypertension in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jianguo He, Chief of Pulmonary Vascular Disease Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2016YFC1304401A
Record Dates: First submitted 2017-06-10; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: COPD; Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — serum and blood cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pulmonary hypertension is a common complication of chronic obstructive pulmonary disease (COPD). It is reported that over half of COPD patients develop pulmonary hypertension. COPD and pulmonary hypertension may have pathological or genetics interactions so that patients having both disorders tend to have poor prognosis. Echocardiography is widely used to detect pulmonary hypertension, but it's not accurate enough. Therefore, high-quality data reflecting the prevalence, disease course and outcome of pulmonary hypertension in COPD is very limited in China. The aim of the study is to detect pulmonary hypertension with right heart catheterization, describe its outcome in Chinese COPD patients and explore the underlying interaction mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Stable chronic obstructive pulmonary disease (COPD) patients

Exclusion Criteria:

* Patients with other serious respiratory diseases
* Patients with pulmonary hypertension other than group 3
* Patients with right heart hypertrophy or dysfunction not caused by chronic obstructive pulmonary diseases
* Patients with limited life expectancy
* Patients with history of tracheal intubation or stoke, acute coronary syndrome in 6 months
* Psychopath or addict

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 1708 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
COPD exacerbations | 3 years
  total hospitalizations times due to COPD exacerbations

SECONDARY OUTCOMES:
modified British medical research council (mMRC) score | 3 years
  COPD symptom score
COPD Assessment Test (CAT) score | 3 years
  COPD symptom score
6 minutes walk distance | 3 years
  meters
transplant-free survival rate | 3 years
  transplant-free survival rate in %

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided